CLINICAL TRIAL: NCT05004909
Title: Effectivity of 1 Finger Tip Unit Compared to 2 Finger Tip Units 0.05% Tretinoin Cream Before and After 30% Trichloroacetic Acid Chemical Peeling on Aging Skin
Brief Title: Effectivity of 1 Finger Tip Unit Compared to 2 Finger Tip Units 0.05% Tretinoin Cream
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Irma Bernadette S. Sitohang, MD, PhD - Head of Cosmetic Dermatology Division, Department of Dermatology and Venereology, Faculty of Medicine, Universitas Indonesia, dr. Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TretandTCAPeeling
Record Dates: First submitted 2021-07-27; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Photoaging
Keywords: Photoaging; Tretinoin; Trichloroacetic Acid; Chemical Peeling
MeSH Terms: interventions — Tretinoin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 Fingertip Unit 0.05% Tretinoin (Active Comparator): Subjects were randomized to receive the instructions to use 1 fingertip unit of 0.05% tretinoin cream for 2 weeks before the first chemical peeling. After that, this therapy is instructed to be used for 4 weeks after the chemical peeling procedure with 30% trichloroacetic acid until the scheduled evaluation.
  Interventions: Drug: 0.05% Tretinoin
- 2 Fingertip Units 0.05% Tretinoin (Experimental): Subjects were randomized to receive the instructions to use 2 fingertip units of 0.05% tretinoin cream for 2 weeks before the first chemical peeling. After that, this therapy is instructed to be used for 4 weeks after the chemical peeling procedure with 30% trichloroacetic acid until the scheduled evaluation.
  Interventions: Drug: 0.05% Tretinoin

INTERVENTIONS:
Drug: 0.05% Tretinoin — Topical 0.05% tretinoin cream applied daily every night by the subjects according to assigned randomization

SUMMARY:
This clinical study will compare the efficacy of using one fingertip unit and two fingertip units of 0.05% before and after 30% trichloroacetic acid chemical peel procedure for facial skin rejuvenation in 35-60 years old female patients with Glogau II-III skin classification.

DETAILED DESCRIPTION:
This study is an experimental study with a randomized controlled trial (RCT) design on patients who met the inclusion criteria. Group A will receive pretreatment in the form of 0.05% tretinoin cream which is used as much as one fingertip unit every night, and group B will receive the same cream which should be used as much as two fingertip units. This cream will be used for two weeks before the patients receive a chemical peeling therapy using 30% trichloroacetic acid. The results of therapy will mainly be assessed based on the Dermoscopic Photoaging Scale (DPAS), as well as visual analog scale (VAS) for subjective symptoms and Clinician Erythema Assessment Scale (CEA) for erythema.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 35-60 years old
* Patients with Glogau II-III skin classification
* Patients are willing to participate in the study and sign an informed consent form

Exclusion Criteria:

* Patients with hypertrophic scars or keloid on the face
* Patients with open wound or infection on the face
* History of other topical treatment on the face within 1 month of enrollment
* Pregnant or breastfeeding mother
* Patients and/or their families are not willing to participate in the study.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of Photoaged Skin Condition | Baseline(pre-chemical peeling procedure), immediately after chemical peeling procedure, and 4 weeks after chemical peeling procedure
  using dermoscopic photoaging scale (DPAS). This DPAS assessment is based on yes or no rules on 11 criteria in four facial regions, namely left malar, right malar, forehead, and chin. The criteria were yellowish discoloration, white line, lentigo, hypo- and hyper-pigmented macules, telangiectasia, yellow papules, actinic keratosis, senile comedones, deep wrinkle, superficial wrinkle, and criss-cross wrinkle. Score range is 0-44 points.
Change of Subjective Pain Evaluation | Baseline(pre-chemical peeling procedure), immediately after chemical peeling procedure, and 4 weeks after chemical peeling procedure
  using Visual Analog Scale (VAS). Scale range is 0-10, 0 indicates no pain and 10 indicates severe pain
Change of Erythema Degree | Baseline(pre-chemical peeling procedure), immediately after chemical peeling procedure, and 4 weeks after chemical peeling procedure
  using Clinician Erythema Assessment Scale (CEA). Scale range is 0-4, 0 indicates no erythema and 4 indicates severe erythema
Change in Skin Thickness | Baseline(pre-chemical peeling procedure) and 4 weeks after chemical peeling procedure
  Evaluation with USG of epidermal and dermal layer (in pixels)

CONTACTS AND LOCATIONS:
Overall Officials: Irma BS Sitohang, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Indonesia dr. Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No